CLINICAL TRIAL: NCT06105905
Title: Reducing Reproductive Health Disparities Among Latino Youth Living in Rural Communities
Brief Title: Latino Teen Pregnancy Prevention K23
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Romina Barral, Associate Professor of Pediatrics, UMKC School of Medicine; Research Assistant Professor of Pediatrics, University of Kansas Medical Center; Faculty, Division of Adolescent Medicine, Children's Mercy Hospital Kansas City, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002128; 1K23HD109464-01 (NIH)
Record Dates: First submitted 2023-10-12; First posted 2023-10-30 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy in Adolescence; Rural Health; Hispanic or Latino

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm pilot trial (Experimental): The developed intervention will be delivered in a workshop format by facilitators, over 8 sessions for teens and parent/guardian(s). Feedback will be elicited on delivery mode (virtual, in-person, or hybrid) during the co-development sessions. If in-person/hybrid is suggested, feedback will be elicited about preferred location (e.g., a local community center, sports club, etc.). Sessions will be hosted in either Spanish or English depending on participants' preference, using video conference tools. Teens and parent/guardian(s) will complete a 20-minute survey pre-intervention, immediately after the 8 session intervention, three-month post-intervention, six-month post-intervention, and twelve-month post-intervention. Surveys will assess acceptability and risk behaviors. As in the published Cuidate trials, previously used measures will be used to document validity and comparability.
  Interventions: Behavioral: Healthy futures ("Futuros Saludables")

INTERVENTIONS:
Behavioral: Healthy futures ("Futuros Saludables") — The developed intervention will be delivered in a workshop format by facilitators, over 8 sessions for teens and parent/guardian(s). Feedback on delivery mode (virtual, in-person, or hybrid) during the co-development sessions. If in-person/hybrid is suggested, feedback will be elicited about preferred location (e.g., a local community center, sports club, etc.). Participants will complete sessions, in either Spanish or English depending on participants' preference, using video conference tools. After the delivery of the intervention, facilitators will take field notes and complete a debriefing questionnaire to assess practicality and fidelity. Teens and parent/guardian(s) will complete a 20-minute survey pre-intervention, immediately post-intervention, three-month, six-month, and twelve-month post-intervention. Surveys will assess acceptability and risk behaviors.

SUMMARY:
The study will utilize an exploratory study design, applying formative research methods to inform the development and pilot testing of an unintended teen pregnancy prevention intervention.

DETAILED DESCRIPTION:
The study uses questionnaires and interviews with youth and community members, to co-develop and pilot test an unintended teen pregnancy prevention intervention in an emerging immigrant Latino rural community, aiming to decrease reproductive health disparities in marginalized communities across the country. To achieve this objective, the team will conduct interviews and co-development sessions, to ensure input from key stakeholders in the community, when developing an intervention.

Delineation of Activities:

Research Activities

• Aim 1: Through stakeholder-engaged research, the team will identify key factors (at multiple levels of influence as defined by NIMHD) needed for the co-development of an acceptable and effective teen pregnancy prevention intervention for rural Latino teens: The team will conduct up to 60 key informant interviews to identify barriers to and facilitators of teen pregnancy prevention programming, such as cultural and social norms. Participants will complete a survey to collect demographic data before participating in the interview. Interviews will last 45 to 60 minutes, in either Spanish or English depending on participants' preference, and will be done using video conference tools at the interviewee's location and times of preference to accommodate participants' schedules.

• Aim 2: Using the transcreation framework, co-develop with community partners a teen pregnancy prevention intervention that best fits the community's unique needs and context: Up to 50 key stakeholders will participate in approximately 8 co-development hybrid sessions to discuss, draft, and redraft each module of the Cuidate intervention syllabus, interactive course materials, and activities. The goal of the workgroup is to discuss recommendations and unique needs of local Latino teens (Specific Aim 1) and modify Cuidate in response to local insights. These sessions will be facilitated by the study research team in either Spanish or English depending on the participants' preference. The sessions will be done using a hybrid method that could include in-person interactions and/or video conference tools at the interviewee's location and times of preference to accommodate participants' schedules. Virtual co-development sessions will be conducted via Microsoft Teams. University of Kansas (KU) will utilize Zoom as an alternative option for virtual meetings. In that instance, KU will initiate the Zoom call. In-person, interviews may be conducted at a local church, and/or at a location managed by a Juntos Community Health Specialists.

• Aim 3: Conduct a pilot study to evaluate the feasibility of a co-created teen pregnancy prevention intervention in target Latino rural communities: The co-developed intervention will be delivered in a workshop format by facilitators, over 8 sessions for teens and parent/guardian(s). Feedback on delivery mode (virtual, in-person, or hybrid) will be elicited during the co-development sessions. If in-person/hybrid is suggested, information will be collected about preferred location (e.g., a local community center, sports club, etc.). Participants will complete sessions, in either Spanish or English depending on participants' preference, using video conference tools. After the delivery of the intervention, facilitators will take field notes and complete a debriefing questionnaire to assess practicality and fidelity. Teens and parent/guardian(s) will complete a 20-minute survey pre-intervention, immediately post-intervention, three-month post-intervention, six-month post-intervention, and twelve-month post-intervention (computer-assisted, self-administered, online via Research Electronic Data Capture - REDCap). Surveys will assess acceptability and risk behaviors. As in the published Cuidate trials, previously used measures will be used to document validity and comparability. Surveys will be de-identified; participants will create a code to match surveys without using identifying data.

Those currently enrolled are only from non-trial aims in this module.

ELIGIBILITY:
Inclusion Criteria:

* 14-18 years old,
* speak English or Spanish,
* Parents/LARs.

Exclusion Criteria:

* non-English or non-Spanish speaking
* developmental delayed
* have significant behavioral health issues which may interfere with study participation
* incarcerated minors
* minors in foster care.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
A survey analysis of participant degree of acceptance of conducted intervention using a Likert Scale. | Immediately after intervention
  This outcome measure identifies the degree in which the intervention is accepted by the participant. Acceptability refers to the extent at which the intervention is perceived as agreeable, or satisfactory to the participant. Acceptability is measured using a Likert Scale in a survey immediately after the 8 session intervention is administered. The Likert Scale ranges from 1-4: 1) Newly Approved Intervention Meets my approval, 2) Newly Approved Intervention is appealing to me, 3) I like the Newly Approved Intervention, 4) I welcome the Newly Approved Intervention.
A survey to determine the participants perception of intervention applicability of conducted intervention using a Likert Scale. | Immediately after intervention.
  This outcome measure identifies the extent in which a participant assesses the appropriateness of the conducted intervention. Appropriateness refers to the perceived ft, relevance, or compatibility of the innovation for a given practice setting, provider, or consumer; and/or perceived ft of the innovation to address a particular issue or problem. Appropriateness is measured using a Likert Scale in a survey immediately after the 2-day intervention is administered. The Likert Scale ranges from 1-4: 1) Newly Approved Intervention seems fitting, 2) Newly Approved Intervention seems suitable, 3) Newly Approved Intervention seems applicable, 4) Newly Approved Intervention seems like a good match.
A survey to determine the facilitators perception of the difficulty of implementing the intervention. | Facilitator surveys will occur immediately post intervention. Field notes will be collected during the delivery of the intervention.
  This outcome measure identifies the feasibility for facilitators to conduct the intervention. Feasibility refers to the extent to which an innovation "can be success- fully used or carried out within a given agency or setting". Feasibility will be measured using the facilitator survey that employs a Likert Scale. The Likert Scale ranges from 1-4: 1) Newly Approved Intervention seems implementable, 2) Newly Approved Intervention seems doable, 3) Newly Approved seems easy to use. Feasibility will also be measured using ethnographic field notes that are analyzed using inductively using a grounded theory approach. Weekly meetings will allow for resolution of discrepancies and to establish inter-rater reliability.

SECONDARY OUTCOMES:
A survey analysis of teen sexual behavior risk pre and post intervention. | Average of 20-minute survey pre-intervention, immediately after intervention, three-month, six-month, and twelve-month post-intervention
  This outcome measure analyzes teens' sexual behaviors, to determine their overall sexual risk. The outcome measure analyzes participant condom usage and multiple partners as identities of risk over the last 90 days. The survey is designed to identify if sexual risk is decreased post-intervention for participants (Increase in condom usage and decrease in the number of sexual partners).
A survey analysis of teen sexual intention pre and post intervention. | Average of 20-minute survey pre-intervention, immediately after intervention, three-month, six-month, and twelve-month post-intervention
  The survey will analyze the following: "Attitudes towards protection, Attitudes towards risky behavior, Knowledge of pregnancy risk, Knowledge of sexually transmitted infections risk, Motivation to delay childbearing, Intention measures, Refusal skills, condom negotiation skills". This survey aims to examine if sexual intentions and knowledge have changed between pre and post intervention.
Pregnancy risk/prevention self-efficacy | Average of 20-minute survey pre-intervention, immediately after intervention, three-month, six-month, and twelve-month post-intervention
  Survey analysis of "history of teen pregnancy" and "pregnancy prevention self -efficacy". This survey aims to examine if history of teen pregnancy and self-efficacy in preventing pregnancy have changed between pre and post intervention.
Cultural Pride | Average of 20-minute survey pre-intervention, immediately after intervention, three-month, six-month, and twelve-month post-intervention
  A survey analysis of teen and adult Latino cultural pride. The survey will analyze the following: "Cultural pride and Family interactions" This survey aims to examine the extent of the individual's pride in Latino background and participation in family activities that reflect Latino values and if changes from pre to post intervention.
For teens Healthy Relationships | Average of 20-minute survey pre-intervention, immediately after intervention, three-month, six-month, and twelve-month post-intervention
  The survey will analyze "teen knowledge of healthy relationships" and "communication with parents about healthy relationships" . This survey aims to examine if teen knowledge of healthy relationships and their communication with parents about healthy relationships changes from pre to post intervention.
For Adults difficult conversations | Average of 20-minute survey pre-intervention, immediately after intervention, three-month, six-month, and twelve-month post-intervention
  The survey will analyze the following: " Difficult conversations". This survey aims to examine if parent's perceived competence and self-efficacy to approach difficult conversations with their teen changes from pre to post intervention.
Family Connections | Average of 20-minute survey pre-intervention, immediately after intervention, three-month, six-month, and twelve-month post-intervention
  A survey analysis of motivation to interact with their teen/adult. The survey will analyze the following: "Family connections". This survey aims to examine change in knowledge, attitudes and intentions about interaction with their teen/adult from pre to post intervention.
Communication | Average of 20-minute survey pre-intervention, immediately after intervention, three-month, six-month, and twelve-month post-intervention
  A survey analysis of parent/teen attachment. The survey will analyze the following "parent-teen relationship". This survey aims to examine if there is a change in general parent/teen attachment pre and post intervention.
Mental health: Parent Adolescent Communication scale | Average of 20-minute survey pre-intervention, immediately after intervention, three-month, six-month, and twelve-month post-intervention
  The Parent-Adolescent Communication Scale (PACS) is a measure used to evaluate the quality of communication between parents and adolescents. The measure consists of two subscales, the Open Family Communication subscale, which addresses the degree of openness in communication, and the Problems in Family Communication subscale, which addresses difficulties in communication. This survey aims to examine if there is a change in parent-teen communication about mental health pre and post intervention.
Health care utilization and access | Average of 20-minute survey pre-intervention, immediately after intervention, three-month, six-month, and twelve-month post-intervention
  A survey analysis of healthcare utilization. The survey will analyze if participants have received care in the past 3 months and the type of care received. This survey aims to examine if there is a change in healthcare use and access to health care in general, and in particular for mental and sexual health, pre and post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Romina L Barral, M.D., Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Childrens Mercy Hospital and Clinics, Kansas City, Missouri, United States